CLINICAL TRIAL: NCT01903304
Title: Immunological Impact of High Olive Oil Consumption
Acronym: OOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Simin Meydani, Principal Investigator, Tufts University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FRGN64
Record Dates: First submitted 2011-12-04; First posted 2013-07-19 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Immune Factors
Keywords: Olive oil; DTH; elderly
MeSH Terms: interventions — Olive Oil

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- olive oil (Experimental): intervention with olive oil for 3 months
  Interventions: Other: Olive Oil
- Placebo (Placebo Comparator): Intervention with placebo for 3 months
  Interventions: Other: Olive Oil

INTERVENTIONS:
Other: Olive Oil — 3 months intervention

SUMMARY:
This is a prospective, randomized controlled nutrition intervention trial to determine immunological impact of high olive oil consumption in elderly. Aging is associated with impaired immune response which contributes to higher incidence of infections in elderly. Previously the investigators have shown that the type of fatty acids in the diet influences the immune response. In particular, reducing consumption of fats high in n-6 fatty acids has been shown to improve the immune response in aged. Very few studies have evaluated the role of olive oil, the main oil consumed as part of the Mediterranean diet on the immune response of elderly. The investigators hypothesize that high olive oil consumption will improve immune function in elderly. In addition, the investigators will investigate the effect of high olive oil consumption on gene expression of relevant pathways in circulating mononuclear cells, as well as on cognitive function.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled nutrition intervention trial to determine immunological impact of high olive oil consumption in elderly. Aging is associated with impaired immune response which contributes to higher incidence of infections in elderly. Previously we have shown that the type of fatty acids in the diet influences the immune response. In particular, reducing consumption of fats high in n-6 fatty acids has been shown to improve the immune response in aged. Very few studies have evaluated the role of olive oil, the main oil consumed as part of the Mediterranean diet on the immune response of elderly. We hypothesize that high olive oil consumption will improve immune function in elderly. In addition, we will investigate the effect of high olive oil consumption on gene expression of relevant pathways in circulating mononuclear cells, as well as on cognitive function.

Subject recruitment and enrollment will be conducted at the USDA HNRCA. Following screening, 40 eligible overweight or obese participants aged 65 and above will be randomized into one of two nutrition intervention groups for a period of 12 weeks: [1] Control Typical American Diet A, (N=20) and [2] Experimental Diet B (N=20).

Participants on the Control Diet A will be consuming a low-fiber, high-fat typical American Diet. Those on Diet B will consume a similar diet as the typical American diet, but they will be asked to replace their oil intake with extra virgin olive oil. Dietary counseling will be provided by the study dietitian at the Metabolic Research Kitchen of the Jean Mayer USDA Human Nutrition Research Center on Aging (HNRCA) at Tufts University on where the study oils will be replacing oils in the subjects' diets. Subjects will be followed regularly by the study dietitian throughout the intervention period to provide support and ensure compliance to study protocol. Data collection will take place at baseline, and after the subjects have been on the study diets for a period of three months. Data collection for the study outcome measures of interest will comprise blood drawing, anthropometric measurements, and cellular and immune factors. Specifically, measures will include:

1. in vivo indices of T cell-mediated function [delayed type hypersensitivity (DTH)],
2. plasma inflammation markers (such as IL-1b, IL-6, TNF-a, CRP, MCP-1, sICAM-1, and sVCAM-1),
3. ability of T cells and their subsets (such as CD4 and CD8, naïve and memory) to proliferate,
4. Ex vivo production cytokines and PGE2 by immune cells.
5. Gene expression of relevant pathways using transcriptomics analysis in circulating mononuclear cells.
6. The CANTAB (Cambridge Cognition Ltd, Tunbridge Court, Tunbridge Lane, Bottisham, Cambridge, CB25 9TU, UK) is a computerized cognitive assessment, and
7. Beck Depression Inventory.

This study will be conducted by the Nutritional Immunology Lab, with Dr. Simin Meydani as the PI and Drs. Barnett (Project director), Wu (Lab Director), Dallal (Biostatistician), Saltzman (Study Physician), Sen, Scott, and Ordovas as Co-Investigators. Dr. Ascension Marcos of the Scientific National Research Council (CSIC) is also a Co-I of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Must be willing to be randomized into study groups.
2. Men and women ≥ 65 years of age.
3. Body mass index (BMI) between 25 - 35 kg/m2.
4. Consumption of typical American diet.
5. Must be willing to stop taking multivitamins, and supplements (with the exception of vitamin D and calcium), including fish oil or n-3 fatty acids and herbal supplements, for 30 days prior to and during study participation, if currently taking these.

Exclusion Criteria:

1. Using olive oil or canola oil as the predominant oil for cooking for the past 6 months, but eligible if willing to stop taking these oils for 30 days prior to participation.
2. Currently on a vegetarian diet.
3. Eats more than 3 meals per week at a restaurant.
4. Consumes fish more than three times per week; but eligible if willing to stop fish consumption 30 days prior to participation and during participation..
5. Disordered eating habits:

   * "Crash" diets
   * Bingeing or food sprees
   * Failure to consume a consistent diet, or demonstrates regular changes in patterns of dietary intake.
6. Heavy consumption of alcohol (more than 2 glasses of alcoholic drinks per day).
7. HIV+ by self-report.
8. Autoimmune disease, Type 1 diabetes, celiac disease, inflammatory bowel disease (IBD), multiple sclerosis, rheumatoid arthritis, autoimmune hepatitis.
9. Diseases that impact the immune response such as cancer, except for non-melanoma skin cancer, and other neo-plastic diseases.
10. Chemotherapy, anti-neo plastic or immunosuppressive drugs.
11. Any major illnesses that are uncontrolled (not stable on medication) - uncontrolled liver disease, uncontrolled heart or cardiovascular disease, uncontrolled Hypertension, uncontrolled renal disease, uncontrolled asthma.
12. History of smoking or use of nicotine containing products in the past 6 months.
13. Active infection within 4 weeks of study enrollment, blood draws or skin tests; however, may participate if admission is postponed or rescheduled > 4 weeks after resolution of symptoms.
14. FLU vaccination within 2 weeks prior to study blood draws and skin tests.
15. Currently on antibiotics; if on antibiotics need to be off antibiotics for at least 2 weeks before study enrollment, and 2 weeks prior to blood draws up to 48 hrs after DTH implant (i.e. after second reading). .
16. Chronic prophylactic antibiotic treatment or long term antibiotics.
17. Diagnosis of infections at base¬line will not exclude a subject, but will postpone en¬rollment to 4 wks after symptoms have cleared.
18. Participation in weight reduction program within 6 months prior to study enrollment; but include if enrolled in weight loss program to maintain body weight.
19. History of splenectomy
20. On dialysis
21. Conditions or medications associated with maldigestion or malabsorption, including but not limited to (in the opinion of the study physician), inflammatory bowel disease, chronic pancreatitis, celiac disease, resection of the small intestine, gastric bypass or other surgery for weight loss, and use of orlistat.
22. Known poor compliance to dietary intervention (based on dietary screening interview).
23. Unwillingness to maintain current body weight and level of physical activity during the study period.
24. Consumption of herbal supplements. Interested eligible participants on herbal supplements will be asked to stop taking these while on the study after a 30 day washout period.
25. Use of aspirin, non-steroidal anti-inflammatory medications (NSAIDs) or antihistamine prescribed by a physician or clinician, or the inability to discontinue the use of these substances for 72 hrs before first day blood draw until 48 hrs after DTH implant (i.e. after second reading).

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change in delayed hypersensitivity skin-test (DTH) | baseline and month 3
  Subjects will be tested for the DTH skin response to 3 antigens (tricophyton, tetanus, and candida, plus saline as control) at baseline and 3-mo after supplementation.

SECONDARY OUTCOMES:
change in plasma inflammation markers | Baseline and month 3
  Blood will be collected at baseline and 3-mo after supplementation to determine IL-1b, IL-6, TNF-a, CRP, MCP-1, sICAM-1, and sVCAM-1 levels in the plasma, which provide an in vivo status of inflammation associated with metabolic syndrome

OTHER OUTCOMES:
change in ability of T cells and their subsets (such as CD4 and CD8, naïve and memory) to proliferate | baseline and month 3
  Blood will be collected at baseline and 3-mo after supplementation and peripheral blood mononuclear cells (PBMC) will be isolated. PBMC will be labeled with the tracking dye CFSE and stimulated for 3 days. The cells will be labeled with appropriate antibodies to identify the sub-populations of T cells (CD4 and CD8, naïve and memory) and combined with CFSE tracking, proliferation profile of each sub-population will be obtained.
change in ex vivo production of cytokines and PGE2 by immune cells | baseline and month 3
  Blood will be collected at day 1 and day 2 (duplicate sampling to counter day to day variation in this type of assays) of both baseline and 3-mo after supplementation. Whole blood culture will be stimulated to determine the ability of T cells to proliferate and of immune cells to produce cytokines and PGE2.
change in gene expression of relevant pathways using transcriptomics analysis in circulating mononuclear cells. | baseline and month 3
  Five milliliters blood samples will be collected in the fasting state both at baseline and following 3 months of dietary intervention. Total RNA from mononuclear cells will be isolated and processed to Biotin labeled cRNA at the Nutritional Genomics Lab, JM HNRCA at Tufts University. We will use the GenMapp 2.1 and MappFinder 2.0 software package (www.GenMapp.org) for the Gene Ontology (GO) and pathway analysis.
change in cognitive function using the CANTAB (Cambridge Cognition Ltd, Tunbridge Court, Tunbridge Lane, Bottisham, Cambridge, CB25 9TU, UK) computerized cognitive assessment tool. | baseline and month 3
  We have chosen the following CANTAB modules to assess attention, memory, language and executive function.
change in measure using Beck Depression Inventory | baseline and month 3
  At baseline and the 3 month follow-up, participants will be tested for cognitive function and will be administered the Beck Depression Inventory - II.

CONTACTS AND LOCATIONS:
Overall Officials: Simin N Meydani, DVM, PhD, Principal Investigator — Human Nutrition Research Center on Aging; Junaidah B Barnett, MCH(N), PhD, Study Director — Human Nutrition Research Center on Aging
Locations (1):
- Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Background] Rozati M, Barnett J, Wu D, Handelman G, Saltzman E, Wilson T, Li L, Wang J, Marcos A, Ordovas JM, Lee YC, Meydani M, Meydani SN. Cardio-metabolic and immunological impacts of extra virgin olive oil consumption in overweight and obese older adults: a randomized controlled trial. Nutr Metab (Lond). 2015 Aug 7;12:28. doi: 10.1186/s12986-015-0022-5. eCollection 2015. PMID 26251666